CLINICAL TRIAL: NCT03822923
Title: Effects of Neurodynamics on Spasticity in Upper Extremity of Stroke Patients.
Brief Title: Neurodynamics on Spasticity in Upper Extremity of Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIU Nafeesa Zamurd
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Stroke
Keywords: Neurodynamics; Spasticity; Stroke
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Neurodynamics (Dynamic Neural Mobilization) with conventional treatment (stretching, AROM) will be applied.
  Interventions: Other: Experimental group
- control group (Active Comparator): Conventional treatment (stretching, AROM) will be applied
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental group — Neurodynamics with conventional treatment. Intervention will be applied for 6 weeks (10 reps per set, 1 set per day, 3 days per week) for 30 minutes
  Arms: Experimental group
Other: Control group — Conventional treatment
  Arms: control group

SUMMARY:
Data will be collected from 40 patients with hemiplegia, caused by stroke from DHQ hospital Jhelum. its an RCT Neurodynamics with conventional treatment to experimental group and conventional treatment alone to control group will be applied for 6 weeks.

Simple random sampling will be done and randomization will be done through tossing a coin. Intervention wil be applied and assesment will be done through fugl-meyer upper extremity scale, Modified Aashwarth scale,goniometry and action research arm test at zero, 3rd and 6th week.

DETAILED DESCRIPTION:
Informed consent was taken and patients were assessed for eligibility and patients who meet the inclusion criteria were randomized through simple random sampling into experimental and control group. Zero, 3rd and 6th week assessment was done through Action research arm test to assess upper limb performance, Goniometry to assess range of motion, Fugl-meyer upper extremity scale FMUE to assess motor functioning, sensation and joint functioning and modified ashworth scale MAS to assess spasticity. Intervention was applied for 6 weeks. The intervention in control group (n=23) was conventional treatment which includes stretching (static stretching for 20 sec) and range of motion exercises (within limit of range) . Intervention was administered one set per day (12 reps per set) four repetitions for each movement direction for 3 days a week, over a course of 6 weeks.

The intervention in experimental group (n=23) was conventional treatment which includes stretching (static stretching for 20 sec) and range of motion exercises (within limit of range) with neurodynamics (Dynamic neural mobilization technique) which includes median, ulnar and radial nerve mobilization. Peripheral nerve was stretched for 20 sec with addition of dynamic movement which was performed after every 2 sec for a total of 20 sec. Neurodynamics was administered, one set per day (10 rep per set) , for 3 days a week, over a course of 6 weeks. Normality of data was checked through shapiro wilk test as sample size is <50 and parametric or non-parametric tests were applied accordingly through SPSS version 21.

Rhythmic neurodynamics accelerated the nerve conduction velocity more than the general neurodynamics. Positive effect of neurodynamics to reduce tone, increase range and improve function of stroke patients were determined in 2016. Combination of neural mobilization and Botulinum toxin-A is effective to reduce pain and increase ranges of motion.Decrease in anxiety also occurs. Botulinum toxin inhibits release of acetylcholine causing a blockade of the neuromuscular patches without affecting the antagonist muscles resulting in reduced spasticity.

Neural mobilization is effective than conventional neural mobilization to increase β-waves and decrease μ-rhythms in C3 and C4 areas of cerebral cortex (primary motor areas). Neural mobilization was effective for improving range of motion of shoulder joint in all degree of freedom by reducing muscle tension and increasing extensibility of neural tissue. Neural mobilization is effective to reduce spasticity in bicep brachii muscle. Decrease in myoelectric activity is the mechanism behind reduction of tone in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Modified Ashworth scale (MAS) of 1 to 3, chronic cases (6 -12 months)

Exclusion Criteria:

* Modified Ashworth scale (MAS) 0 and 4, painfull upper extremity, orthopedic problem (e.g fracture)
* In upper extremity, UMNL other than stroke,
* Any signs of inflammation, infection or malignancy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Modified Ashwarth Scale | 6th weeks
  Effects of neurodynamics to reduce spasticity in uppper extremity will be assesed through Modified Ashwarth Scale changes from Baseline. Modified Ashwarth Scale is a specific scale to asses spasticity. Scoring is done from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension).

SECONDARY OUTCOMES:
Range of motion Shoulder Joint (Flexion, Extension, abduction, internal rotation, external rotation ) | 6th weeks
  Changes from the baseline. Range of Motion of Shoulder will be Assess through Goniometer.
Fugl Meyer upper extremity scale | 6th weeks
  Changes from the Baseline. Fugl Meyer is a stroke specific, performance based impairment index designed to assess motor functioning, sensation and joint functioning. The FMUE Scale comprises 33 items, each scored on a scale of 0 to 2, where 0 = cannot perform, 1 = performs partially and 2 = performs fully. FMUE Scale scores < 31 corresponded with 'no to poor' upper extremity capacity, while 32 to 47 represented 'limited capacity', 48 to 52 represented 'notable capacity' and 53 to 66 represented 'full' upper extremity capacity.
Action research arm test (ARAT) | 6th week
  Changes from the baseline. Action research arm test is highly reliable and valid 19 items tool (grasp (6 items), grip(4 items), pinch (6 items) and gross movement (3 items) which is used to asses upper extremity performance (coordination, dexterity and functioning). In ARAT scoring is done from 0 (unable to complete) to 3 (complete with normal movement). Scores on the ARAT range from 0-57 points, with a maximum score of 57 points indicating better performance. The ARAT can be used to predict the functional recovery of the upper extremity in stroke rehabilitation. Scores of less than 10 points, between 10-56 points, and 57 points correlate with poor, moderate, and good recovery respectively.
Range of motion of elbow joint ( flexion, extension, forearm Supination , Pronation) | 6th week
  Changes from the baseline. Range of Motion of Elbow joint will be Assess through Goniometer.
Range of motion of Wrist joint (flexion, extension , ulnar deviation , thumb abduction ) | 6th Week
  Changes from the baseline Range of Motion of wrist joint will be Assess through Goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santana AL. Efeito da mobilização neural na amplitude articular do ombro em pacientes acometidos com acidente vascular encefálico. Revista Inspirar: movimento & saúde. 2013; (5)6:7-10.
- [Background] Jeong Kang et al, The Effects of Rhythmic Neurodynamic on the Upper Extremity Nerve Conduction Velocity and the Function for Stroke Patients, JKPT 2017, Volume 29 No. 4.
- [Background] Alan Carlos Nery dos Santos et al, The effects of neural mobilization as a therapeutic option in the treatment of stroke, MTP and Rehab journal 2017, ISSN 2236-5435.
- [Background] Villafane JH, Silva GB, Chiarotto A, Ragusa OL. Botulinum toxin type A combined with neurodynamic mobilization for upper limb spasticity after stroke: a case report. J Chiropr Med. 2012 Sep;11(3):186-91. doi: 10.1016/j.jcm.2012.05.009. PMID 23449315
- [Background] Raid Saleem Al Baradie et al, The effects of Neurodynamics and mobilization in Stroke Rehabilitation- a Systematic Review, Majmaah Journal of Health Sciences 2017, Vol.5, issue 2.